CLINICAL TRIAL: NCT00213070
Title: Double-Blind Trial of Miglitol in Type 2 Diabetic Patients With Insulin Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MG1005
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: alpha-glucosidase inhibitor,Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — miglitol

INTERVENTIONS:
Drug: Miglitol

SUMMARY:
The purpose of this study is evaluate the clinical efficacy and safety of Miglitol in patients with Type2 Diabetes Mellitus with treated insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetes
* Criteria of postprandial plasma glucose and HbA1c are met

Exclusion Criteria:

* Type1 diabetes
* Patients with antidiabetic drugs
* The other exclusion criteria are met

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Promotion Group, Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (16):
- Japan (16):
  - Aichi
  - Chiba
  - Fukuoka
  - Gifu
  - Gunma
  - Hokkaido
  - Ibaraki
  - Kagoshima
  - Kanagawa
  - Kumamoto
  - Miyazaki
  - Okinawa
  - Ōita
  - Saitama
  - Shiga
  - Tokyo